CLINICAL TRIAL: NCT01284764
Title: Efficacy of a Low Volume of Water Intake and Mosapride for Endoscopy Preparation in Gastric Cancer Patients With Subtotal Gastrectomy: A Randomized Controlled Trial
Brief Title: Efficacy Study of a Low Volume of Water Intake and Mosapride for Endoscopy in Patients With Subtotal Gastrectomy
Acronym: SMW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Eun Hee Seo, fellow, Inje University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HGI-2011-01
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Foreign Body Left During Endoscopic Examination
Keywords: Endoscopy; Gastrectomy; Stomach neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — mosapride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- midnight fasting (No Intervention): The patients in this group will have midnight fasting the day before endoscopic examination
- Mosapride, low volume of water (Active Comparator): The patients in this group will take mosapride and a 500mL water at evening of the day before endoscopic examination.
  Interventions: Drug: Mosapride

INTERVENTIONS:
Drug: Mosapride — Mosapride 10mg, one dosage, once evening of the day before the endoscopy
  Other Names: Gasmotin
  Arms: Mosapride, low volume of water

SUMMARY:
A low volume of water intake and mosapride will effectively reduce food residue in remnant stomach for patients who had undergone subtotal gastrectomy due to gastric cancer.

DETAILED DESCRIPTION:
We evaluate that a 500mL of water intake and mosapride will effectively reduce food residue in remnant stomach for patients who had undergone subtotal gastrectomy due to gastric cancer. We plan to compare this method with routine midnight fasting method for endoscopy in patients with subtotal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who had subtotal gastrectomy for gastric cancer

Exclusion Criteria:

* Pregnancy
* Lactation
* History of anastomotic stricture
* Recurrent advanced gastric cancer
* Poor general condition( > 2 ECOG)
* Other disseminated malignancy
* Significant renal failure or congestive heart failure (CHF)
* Liver failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Degrees of food residue using endoscopic scoring system | six months
  We plan to evaluate how much a low volume of water and mosapride, compared with routine fasting, reduse food residue in gastric remnant for endoscopy.

SECONDARY OUTCOMES:
Tolerability of a low volume of water and mosapride | six months
  We plan to evaluate tolerability of a low volume of water and mosapride compared with routine fasting for endoscopy preparation in patients with subtotal gastrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Eun Hee Seo, M.D., Principal Investigator — Haeundae Paik Hospital; Tae Oh Kim, Ph.D., Study Director — Haeundae Paik Hospital
Locations (1):
- Haeundae Paik Hospital, Inje University School of Medicine, Busan, South Korea